CLINICAL TRIAL: NCT01113060
Title: Aspirin Effectiveness in Coronary Artery Disease Patients in Ireland
Brief Title: Aspirin Effectiveness Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Prof Dermot Kenny, Prof. Dermot Kenny, Royal College of Surgeons, Ireland
Other Study IDs: INFACTs2010-001
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Aspirin; Secondary Prevention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAD patients: Representative sample of coronary artery disease patients receiving aspirin therapy for secondary prevention

SUMMARY:
Aspirin is an effective medicine for prevention of heart attacks in patients with coronary artery disease and works by preventing clots from forming. In previous studies aspirin has been found to be ineffective in between 2% and 65% of patients but none of these studies have looked specifically at coronary artery disease patients in Ireland. This study is being done to identify the percentage of patients in Ireland whose aspirin is not working effectively and help identify factors that could be used to target interventions to increase aspirin's effectiveness in Irish patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients with documented coronary artery disease
* Current treatment with any dose of aspirin daily for a minimum of 3 months
* Able to provide written informed consent based on competent mental status

Exclusion Criteria:

* Myocardial infarction, unstable angina or stroke during the preceding three months
* Platelet count <125,000/mm
* Known haematological disorders
* Active malignancy on current chemotherapy or a recent diagnosis of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Representative sample of coronary artery disease patients in Ireland receiving aspririn therapy for secondary prevention of cardiovascular events
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with non-response to aspirin | Following a minimum of 3 months of daily aspirin use
  Prevalence of non-response to aspirin in coronary artery disease patients in Ireland by measurement of serum thromboxane B2

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dermot Kenny, MB, BCh, BAO, MD, Principal Investigator — Royal College of Surgeons, Ireland
Locations (1):
- Beaumont Hospital, Dublin, Dublin, Ireland